CLINICAL TRIAL: NCT01459549
Title: The Role of Roux-en-Y Hepaticojejunostomy in Hepatolithiasis Patients With Sphincter of Oddi Laxity: an Open-label Randomized Controlled Trial
Brief Title: Roux-en-Y Hepaticojejunostomy for Hepatolithiasis With Sphincter of Oddi Laxity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYYYSOL
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Hepatolithiasis; Sphincter of Oddi Dysfunction
Keywords: Hepatolithiasis; Sphincter of Oddi Dysfunction; Roux-en-Y hepaticojejunostomy; randomized controlled trial
MeSH Terms: conditions — Sphincter of Oddi Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): The common bile duct will be maintained for bile drainage in the control arm.
- Trial arm (Experimental): Roux-en-Y hepaticojejunostomy will be performed for bile drainage in the trial arm.
  Interventions: Procedure: Roux-en-Y hepaticojejunostomy

INTERVENTIONS:
Procedure: Roux-en-Y hepaticojejunostomy — All participants received routine perioperative care and followed the same surgical principles: removing affected liver segments, clearing stones, correcting strictures, and then restoring bile drainage. The primary indications for hepatectomy were unilobar or segmental diseases and the presence of the following lesions in the affected liver segment or lobe: 1) multiple stones with biliary strictures that cannot be cured via choledochoscopy, 2) atrophy, fibrosis, and multiple abscesses, and 3) suspicious neoplasia. Biliary exploration was routinely conducted to facilitate stone removal, rectify strictures, and assess the functionality of the Oddi sphincter. Following this, patients would be evaluated for eligibility and assigned accordingly. The sole distinction between the two arms was performing RYHJ or maintaining the common bile duct for bile drainage.
  Arms: Trial arm

SUMMARY:
Objective: Evaluate the role of Roux-en-Y hepaticojejunostomy (RYHJ) in hepatolithiasis patients with sphincter of Oddi laxity (SOL).

Summary Background Data: Hepatolithiasis poses high risks of residual, recurrence, and re-intervention. SOL significantly impacts this condition. RYHJ has been recommended for hepatolithiasis concomitant SOL but without prospective evidence.

Methods: This is an open-label randomized controlled trial recruiting patients with hepatolithiasis concurrent SOL. Patients were randomly assigned (1:1) to undergo RYHJ or not. The primary endpoint was stone occurrence, including residual and recurrence, within a three-year postoperative period. Secondary endpoints incorporated perioperative and long-term outcomes, like episodes of cholangitis and invasive re-interventions for stones and related complications. The analyses followed the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18 and 80 years
2. diagnosed with SOL during operation
3. suitable for a radical surgery including RYHJ
4. hopeful to clear stones via operation or combined with subsequent choledochoscopy
5. provided written informed consent
6. willing to complete a 3-year follow-up

An intraoperative diagnosis of SOL was established if the rhythmic contraction and relaxation of the sphincter of Oddi were not observed under choledochoscope and the flexible choledochoscope (CHF-P20, external diameter, 4.9 mm; Olympus, Tokyo, Japan) could navigate smoothly to the duodenum through the sphincter of Oddi without any pre-dilation interventions.

Exclusion Criteria:

1. with imaging evidences of tumor preoperatively
2. had congenital biliary malformations
3. had ever received biliary operation abandoning the Oddi sphincter, such as choledochoduodenostomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-12-13 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The incidence of stones, including residual and recurrent stones, within three years postoperatively. | A three-year postoperative period
  The term "stone occurrence" pertained to the identification of any bile duct stones with the most reliable imaging modality available during the follow-up period. "Stone residual" described a patient in whom stones were detected during the initial follow-up examination, while "stone recurrence" referred to a patient who exhibited no stones at the first follow-up visit but subsequently presented with stones during later follow-up assessments.

SECONDARY OUTCOMES:
Major complications | perioperation
  Postoperative complications were graded according to the Clavien-Dindo definition and those ranked Grade III or above were defined as major complications. Complications arising during unplanned readmission were also taken into account.
Episodes of cholangitis | 3-year follow-up period
  Episodes of cholangitis, regardless of definite or suspected one. The diagnosis of cholangitis were initially established according to the Tokyo 2007 guidelines and were subsequently revised following the Tokyo 2018 guidelines.
Invasive re-interventions for stones and related complications | 3-year follow-up period
  The term "invasive re-interventions" covered operation, percutaneous transhepatic cholangioscopy, and endoscopic retrograde cholangiopancreatography. The planned choledochoscopy following the initial surgical procedure was not lumped into invasive re-interventions.
Postoperative hospital stays | perioperation
  Hospital stays arising during unplanned readmission were also taken into account
Medical expenses | perioperation
  Medical expenses covered all costs incurred throughout the course, including planned choledochoscopy and unplanned readmissions.
Unplanned readmission within 30 days postoperatively | perioperation

OTHER OUTCOMES:
Cholangiocarcinoma arising | 3-year follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University School of Medicine, Hangzhou, Zhejiang, China